CLINICAL TRIAL: NCT01956656
Title: Efficacy Of Lotus Leaves In Management Of Plaque Induced Gingivitis: A 4 Day Double Blind Clinico-Microbiological Trial.
Brief Title: Efficacy Of Lotus Leaves In Management Of Plaque Induced Gingivitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sri Hasanamba Dental College and Hospital (Other)
Responsible Party: Principal Investigator, Dr.Gopi Kishore.C.R., P.G. student, Sri Hasanamba Dental College and Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: z59p5gy7
Record Dates: First submitted 2013-09-17; First posted 2013-10-08 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Gingivitis
Keywords: lotus leaf, mouthwash, gingivitis
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- lotus leaf mouthwash (Placebo Comparator): 10 ml mouthwash to be used for 4days twice daily
  Interventions: Drug: lotus leaf mouthwash
- placebo mouthwash (Placebo Comparator): 10 ml mouthwash to be used for 4 days twice daily

INTERVENTIONS:
Drug: lotus leaf mouthwash — Saline mouthwash to be used for 4 days twice daily by one group the other group the lotus leaf mouthwash
  Other Names: Lotus mouthwash
  Arms: lotus leaf mouthwash

SUMMARY:
Due to difficulties in maintenance of an effective mechanical oral hygiene regime, effective chemical adjunctive measures will likely significantly contribute to overall oral health, the function of which should be to augment mechanical plaque control. Traditionally, in Chinese medicine the lotus leaf has been used for treating gingival inflammation. An extract of lotus leaves have demonstrated significant antibacterial activity against some of the periodontopathogens.

DETAILED DESCRIPTION:
The objective of the present research is to evaluate the efficacy of a lotus leaf mouth wash in management of plaque induced gingivitis.

Study design: 30 systemically healthy volunteers will be randomly allocated into two arms

Arm A: Lotus leaf mouth wash (aqueous) group [Test group] Arm B: Placebo mouth wash group [Control group]

All the volunteers are instructed to refrain from tooth brushing 24 hours before the examination. Clinical parameters (plaque index, bleeding index and gingival index)will be measured and the plaque samples are collected from subjects from each group for microbiological analysis. All the participants will undergo scaling, and they were instructed to refrain from tooth cleaning procedures and were advised to use the prescribed mouth wash twice daily for 4 days. All volunteers were recalled on 5th day for clinical and microbiological analysis. Statistical analysis and results are awaited

ELIGIBILITY:
Inclusion Criteria:

1. Subjects willing to comply with the study protocol & instruction.
2. Clinically diagnosed with chronic gingivitis.
3. No history of allergies to herbal formulations.
4. No history of periodontal therapy within the previous 6 months.
5. No history of antibiotic therapy within the previous 6 months.

Exclusion Criteria:

1. Any systemic diseases
2. Use of tobacco or tobacco related products
3. Pregnant woman and lactating mothers
4. Subjects that had used any type of antibacterial mouthrinse within 4 weeks of recruitment in to the study.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2013-09; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Plaque induced gingivitis | 4 days
  Gingivitis is measured using, Sillness&Loe(1964):Plaque Index Gingival index(GI)-Loe&Sillness(1963) before and after dispensing of mouthwash.

SECONDARY OUTCOMES:
Grams Staining of the plaque collected from the subjects | 4 days
  Supra-gingival plaque sample are taken microbiological(gram staining)analysis before and after mouthwash dispensing.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Ravindra Shivamurthy, MDS, Principal Investigator — Sri Hasanamba Dental College and Hospital
Locations (1):
- Sri Hasanamba Dental College and Hospital, Hassan, Karnataka, India